CLINICAL TRIAL: NCT05790798
Title: The Effect of Occupational Therapy-Based Instrumental Activities of Daily Living Intervention on Stress Level, Quality of Life, and Participation in People With Disabilities
Brief Title: The Effect of Occupational Therapy-Based Instrumental Activities of Daily Living Intervention in People With Disabilities
Acronym: IADLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gokcen Akyurek, Assoc Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59.2023fbu
Record Dates: First submitted 2023-03-16; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Disability Physical
Keywords: Participation; Stress Level; Quality of Life; Instrumental Activities of Daily Living

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The universe of this research, which has a randomized controlled design, is all people with disabilities aged 18 and older who are attended at the Etimesgut Family and Life Center in Ankara. The inclusion criteria of this study were to be 18 years of age or older, to have a score of 17 and below according to the Lawton-Brody Instrumental Activity of Daily Living Scale, to have a score of 24 and above in the Modified Mini-Mental test. In addition, there are some exclusion criteria for research. Exclusion criteria from the study were: Having a communication problem that prevented the participant from completing the assessment and the kits; not participating regularly in the intervention program. For this study, people who attended the Family and Life Center and people with disabilities who regularly come to this center for various reasons were contacted. People (n=35) who met the criteria of the study were informed about the study and invited to participate in this study.
  Interventions: Other: occupational therapy-based instrumental daily living activities intervention
- Control Group (Active Comparator): The universe of this research, which has a randomized controlled design, is all people with disabilities aged 18 and older who are attended at the Etimesgut Family and Life Center in Ankara. The inclusion criteria of this study were to be 18 years of age or older, to have a score of 17 and below according to the Lawton-Brody Instrumental Activity of Daily Living Scale, to have a score of 24 and above in the Modified Mini-Mental test. In addition, there are some exclusion criteria for research. Exclusion criteria from the study were: Having a communication problem that prevented the participant from completing the assessment and the kits; not participating regularly in the intervention program. For this study, people who attended the Family and Life Center and people with disabilities who regularly come to this center for various reasons were contacted. People (n=35) who met the criteria of the study were informed about the study and invited to participate in this study.
  Interventions: Other: Quite recreation activity

INTERVENTIONS:
Other: occupational therapy-based instrumental daily living activities intervention — Occupational therapy-based instrumental activities of daily living intervention were applied to 9 people with disabilities in the intervention group, with sessions consisting of 45 minutes twice a week (totally 8 weeks/16 sessions). While the activity intervention program was being created for the intervention group, the problem areas in the ADL and IADL determined by the evaluations made before the intervention were identified. Ten occupation kits including 2 ADLs (dressing and feeding nutrition), and 8 IADLs (laundry, meal preparation, light cleaning, paperwork, use of technology, lifting and carrying, fine motor and gross motor leisure groups) were used as interventions. Various materials (jar, shirt, spoon, teapot, play dough, stapler, plastic bag, sponge, etc.) were prepared to be used in each occupation kit and to simulate daily activities.
  Arms: intervention group
Other: Quite recreation activity — For the control group, information about the scope, duration and requirements of the research was shared throughout the process. During this period, reading activities continued. The final evaluation of all participants was made at the end of the 8th week of the study and the study was completed.
  Arms: Control Group

SUMMARY:
The aim of this study was to investigate the effects of occupational therapy-based instrumental activities of daily living intervention on stress levels, quality of life, and participation in people with disability. The participants were recruited from the Etimesgut Family and Life Center in Ankara. In this study, an individualized occupational therapy-based instrumental activities of daily living intervention were implemented for a total of 8 weeks, lasting 16 sessions, which included an intervention group (n=9) and a control group (n=9). Changes before and after the intervention were assessed with the Lawton-Brody Instrumental Activities of Daily Living Scale, Waisman Activities of Daily Living Scale, Modified Mini-Mental State Examination Test, SF-36 Health Survey Questionnaire, Perceived Stress Scale, and Community Integration Questionnaire.

DETAILED DESCRIPTION:
The concept of disability refers to the limitation in activity and social participation and loss of function due to the inability to fulfill the roles expected from the people depending on the level of development, sex, and social factors resulting from an impairment or handicap. The number of people with disabilities is increasing daily in the world, and it was determined that 15.6% of the population over 18 has a disability. People with disabilities experience problems in activities such as bathing, dressing, eating, shopping, money management, preparing food, cleaning, and using drugs, due to physical, cognitive, sensory, and psychosocial impairments. The above-mentioned activities are the tasks of everyday life called activities of daily living (ADL). ADLs are classified as basic activities of daily living (basic ADLs; bathing, eating, toilet, etc.), and instrumental activities of daily living (IADLs; shopping, money management, meal preparation, shopping, dog walking, paying bills, etc.).

People with disabilities need IADLs to a large extent in order to continue living more independently in the community. IADLs are meaningful and purposeful activities that give meaning to people's lives and reflect their social values and cultures. IADLs include activities such as taking care of others, using public transport, health management, and household chores, and have a more complex structure than basic ADLs. Unlike basic ADLs, IADLs require more complex cognitive skills such as planning, organization, decision-making, and executive functions, or fine motor, visual sharpness, or hearing skills. In addition, IADLs are also affected by contextual factors (age, sex, habits, education, culture, environment, etc.) independently of daily living activities. Because IADLs are carried out in many social areas outside the home and include activities based on the people's home, work, school, and social participation. Factors such as environmental suitability, social stigma, and stress of people with disabilities, limit participation in their IADLs and negatively affect their quality of life. Therefore, it is seen that low social participation, decreased quality of life, and increased perceived stress are closely related to IADL performance problems.

In the literature, it is seen that intervention methods are used to improve the IADLs of people with disabilities. Clarke et al. implemented an 8-week physiotherapy and occupational therapy-based intervention program in people with mild and moderate Parkinson's disease (n=762). They made individualized practices on sleep, fatigue, personal care, dressing, in-home mobility, housework, and environmental problems within the scope of the intervention. As a result, it was observed that there was a significant increase in IADL performance, and they recommended the use of activity-based intensified intervention programs for future studies. In a survey study conducted with 105 hand therapists in the USA, 97% of therapists stated that interventions that include meaningful and purposeful activities would be more beneficial for people with upper extremity problems, rather than traditional intervention programs using physical agent modalities or progressive resistance exercises. Egan et al. reported a significant increase in the performance and satisfaction levels of self-care, productivity and leisure activities of the therapy group in the activity-based intervention program applied to improve the occupational performance of 16 people with stroke. Studies with high levels of evidence have emphasized that the use of the daily living activities in intervention programs improves the quality of life of people with disabilities. Politis et al. implemented a 4-week kit-based intervention that included activities of daily living for 37 people with dementia. As a result of the intervention, it was found that the increased quality of life and decreased apathy in people with dementia. It has been stated that the use of kits in intervention programs is relatively inexpensive compared to traditional intervention programs, it is colorful and interesting, is enthusiastically welcomed by people, and it is easy to build. In another study, it was determined that 10 activity kits used to improve the leisure activities of people with Alzheimer's and dementia living in nursing homes increased the quality of life of people.

In occupational therapy, Dy and Yancosek, who developed IADLs kits consisting of daily living activities, created an 8-week intervention program within the scope of hand rehabilitation. Activity kits were used to examine the personal opinions of occupational therapists in terms of the ease of application of the kits before and after they were applied to people. As a result, the use of activity kits in evaluation and interventions has been suggested because they are easy and functional compared to biomechanical intervention programs. Berlet and Kaskutas prepared 10 activity kits in the hand therapy clinic for 642 people who have undergone hand surgery, for the areas of basic and instrumental ADLs where they have the most difficulty. They sent the prepared kits to 30 occupational therapists working in the fields of hand and community rehabilitation and received their opinions about these kits. Occupational therapists stated that the kits eliminate the waste of time in building the materials to be used during the intervention and increase the efficiency of the intervention as it deals with the occupational performance of the kits.

In the systematic reviews, it is seen that studies examining the effects of interventions for IADLs are more common in the elderly and that IADL interventions for people with disabilities are limited. In addition, in studies with IADL kits, programs that develop fine motor skills were focused on. According to the studies, it was thought that the proposed IADL interventions to increase the independence of individuals with disabilities should be planned with a new approach. Therefore, it was aimed to examine the effect of the intervention to be made with the kits created for IADLs on people with disabilities. Specifically, The aim of this study was to investigate the effect of occupational therapy-based instrumental activities of daily living intervention on stress levels, quality of life, and participation in people with disabilities.

ELIGIBILITY:
Inclusion Criteria:

* were to be 18 years of age or older,
* to have a score of 17 and below according to the Lawton-Brody Instrumental Activity of Daily Living Scale,
* to have a score of 24 and above in the Modified Mini-Mental test.

Exclusion Criteria:

* not participating regularly in the intervention program.
* Having a communication problem that prevented the participant from completing the assessment and the kits;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Lawton-Brody Instrumental Activities of Daily Living Scale | 8 weeks
  It consists of 8 questions including information about telephone use, meal preparation, shopping, doing daily household chores, laundry, getting on transportation, traveling, medication use and management of finances.

SECONDARY OUTCOMES:
Waisman Activities of Daily Living Scale (W-ADL): | 8 weeks
  It is a scale developed according to the measurement criteria in the literature to measure the ADL of adolescents and adults with developmental disorders (Maenner et al., 2013). It aims to measure the level of independence while performing typical daily living activities in developmental disorders.
Modified Mini-Mental State Examination Test (MMSE-E): | 8 weeks
  It was created by Folstein et al. (1975) with the aim of evaluating the cognitive skills of people. The validity and reliability study were conducted by Babacan et al. (2014) for the Turkish population.
SF-36 Health Survey Questionnaire: | 8 weeks
  The SF-36 assesses quality of life without being specific to any age, disease, or treatment group. It includes 36 questions in eight sub-dimensions: Physical Functioning, Social Functioning, Role Limitations (Physical Problems, Emotional Problems), Vitality, Bodily Pain, General Health Perceptions, and General Mental Health (Ware et al., 1993).
Perceived Stress Scale (PSS): | 8 weeks
  The Perceived Stress Scale (PSS) developed by Cohen et al. (1997). Consisting of 14 items in total, PSS is designed to measure how stressful a person's life is perceived to be. Participants evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)".
Community Integration Questionnaire (CIQ): | 8 weeks
  This questionnaire developed by Willer et al. (1993) to assess community participation. The CIQ consists of 15 questions that assess a person's participation in home and family life, social and productive activities.

CONTACTS AND LOCATIONS:
Overall Officials: Gokcen Akyurek, Phd, Principal Investigator — Assoc Prof
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author, upon reasonable request.